CLINICAL TRIAL: NCT03885661
Title: Vascepa to Accelerate Lipoprotein Uptake and Elimination (VALUE): An Open-Label, Mechanistic, Randomized, Controlled, Single-Center Trial of AMR101 in Patients With Dyslipidemia
Brief Title: Vascepa to Accelerate Lipoprotein Uptake and Elimination
Acronym: VALUE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Amarin Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 823489; AMR-01-01-0024 (Other Grant/Funding Number: Amarin Pharma, Inc.)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Lipid Disorder; Triglycerides High; Dyslipidemias
MeSH Terms: conditions — Lipid Metabolism Disorders; Hypertriglyceridemia; Dyslipidemias | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Intervention Model Description: Parallel, randomized, controlled mechanistic pilot/feasibility experiment focused on elucidating detailed mechanism of action for apolipoprotein turnover kinetics changes using intravenous infusions of stable isotopes in a clinical/translational metabolic unit.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Reference therapy is usual care, so the subject and coordinators are unblinded to assignment, but investigators and outcomes assessors are blinded to assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Icosapent ethyl (Experimental): Icosapent ethyl with a total daily dose of 4 grams, as 2 x 1 gram capsules by mouth twice daily, against a statin background
  Interventions: Drug: Icosapent Ethyl 1000 MG [Vascepa]
- Usual Care (No Intervention): Statin background

INTERVENTIONS:
Drug: Icosapent Ethyl 1000 MG [Vascepa] — Icosapent ethyl is an ethyl ester of the omega-3 fatty acid eicosapentaenoic acid (EPA). The empirical formula of icosapent ethyl is C22H34O2 and the molecular weight is 330.51. The chemical name for icosapent ethyl is ethyl all-cis-5,8,11,14,17-icosapentaenoate.
  Other Names: AMR101
  Arms: Icosapent ethyl

SUMMARY:
This study is a Phase 1 pilot/feasibility mechanistic experiment to help clarify the mechanism of action of an EPA-rich fish oil preparation, icosapent ethyl, on lipid changes in statin-treated patients with residual triglyceridemia.

DETAILED DESCRIPTION:
This is a prospective randomized, controlled pilot/feasibility experiment in a small number of statin-treated patients with residual triglyceridemia assigned to chronic daily exposure to icosapent ethyl 4 g daily vs usual care to get preliminary data to ultimately design a definitive hypothesis-testing experiment to clarify the mechanism of action whereby icosapent ethyl alters lipoprotein kinetics. The formal statistical aim is to develop statistical parameters such as central tendency, dispersion, and distributional shape to design a robust hypothesis-testing study. The primary outcome is based around stable-isotope lipoprotein kinetics, specifically apolipoprotein B kinetics.

ELIGIBILITY:
Inclusion Criteria:

- 1. Triglyceridemia, defined as:

1. statin-treated TG > 200 mg/dL -and/or-
2. statin-treated TG > 150 mg/dL -plus- statin-treated HDL < 45 [men] or < 55 [women] 2. Self-reported Caucasian-majority race, defined as 3 out of 4 grandparents Caucasian 3. Subjects between the ages of 21 and 75 years of age inclusive 4. Ability to understand and agree to informed consent 5. Are reliable and willing to make themselves available for the duration of the study, comply with study procedures, agree not to participate in other clinical experiments, and agree not to donate blood products during the study

   Exclusion Criteria:
   * 1. Diagnosis of idiopathic or otherwise active diabetes: History of resolved gestational or drug-induced diabetes is acceptable, but history Type I or Type II diabetes are exclusionary.

     2. Use of medications indicated for the treatment of diabetes within 6 weeks of the first experimental visit (see Prohibited Treatments) 3. History of a myocardial infarction (MI), unstable angina leading to hospitalization, coronary artery bypass graft surgery (CABG), percutaneous coronary intervention (PCI), uncontrolled cardiac arrhythmia, carotid surgery or stenting, stroke, transient ischemic attack, carotid revascularization, endovascular procedure or surgical intervention within 6 months of baseline.

     4. Known inefficacy to TG-lowering doses of fish oils (e.g. >= 4 caps daily of prescription fish oil or >= 6 caps daily of supplemental fish oil).

     5. TG > 500 mg/dL as the average of valid, statin-treated values 6. BMI > 40 kg/m2 7. BMI < 20 kg/m2 8. Evidence of previously undiagnosed diabetes: Average fasting glucose during screening > 125 mg/dL 9. Known familial lipoprotein lipase impairment or deficiency (Fredrickson Type I), Apo C II deficiency, or familial dysbetalipoproteinemia (Fredrickson Type III).

     10. Severe allergy to fish, unless non-allergic response to fish oil is established (n.b. most fish allergies are to the proteins as opposed to the fats, so with highly-purified oils the risk of a true allergy is remote).

     11. Known intolerance or contraindication to Vascepa, and if the former is unknown, known intolerance or contraindication to fish oil 12. Any surgical or medical condition that may interfere with absorption, distribution, metabolism, or excretion of EPA or DHA.

     13. History of extreme triglyceridemia (TG > 1000 mg/dL) or pancreatitis from triglyceridemia, regardless of whether it is currently controlled.

     14. Medical condition that would prohibit fasting (e.g. diagnosis of insulinoma or postabsorptive hypoglycemia).

     15. Significant disinclination to dairy products (e.g. lactose intolerance, inviolable dietary restrictions). All participants will receive a test dose of the fat challenge during the screening visit, which consists of heavy cream and lactase enzyme. Many people with lactose intolerance successfully avert symptoms by correcting their lactase deficiency with lactase supplements. We will allow these people to participate because we will allow them to take their preferred brand and dose of lactase supplement beyond the lactase in the fat challenge if needed. However, we still require that they are able to tolerate the test dose given during screening.

     16. History of a non-skin malignancy within the previous 5 years. 17. Uncontrolled thyroid disease. 18. Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition.

     19. Major surgery within the previous 6 weeks. 20. Subjects who have undergone any organ transplant. 21. History of illicit drug use within the past 3 years, or regular alcohol use of greater than 14 drinks per week. For clarity, illicit substances are per Federal law or regulations in effect at the time of first approval of this protocol.

     22. Women who are breast-feeding. 23. Women of childbearing potential must have a negative urine pregnancy test at screening and baseline visits and be willing to have additional urine pregnancy tests during the study.

     24. Sexually active subjects (both women and men) must be willing to use a medically accepted method of contraception from screening visit until month after last dose of study drug 25. Significant or unstable medical or psychological conditions, including known or suspected personality disorders, that could compromise the subject's safety or successful participation in the study in the opinion of the investigator.

     26. Subject-reported history of HIV and/or use of HIV medications 27. History of symptomatic gallstone disease unless definitively treated (e.g. condition successfully treated with cholecystectomy without recurrent or residual biliary disease).

     28. History of bariatric surgery or other major gastrointestinal surgery associated with major disruptions to drug absorption.

     29. Anticipation of major surgery during the screening or treatment periods of the study 30. Participants with the following conditions will opt out of heparin exposure for lipase determinations, but will be allowed to participate in the overall protocol.

     31. History of intolerance or adverse reaction to therapeutic or sub-therapeutic heparin regimens 32. History of intracerebral hemorrhage 33. History of significant GI bleed, unless definitively treated without recurrence 34. Women with dysfunctional uterine bleeding 35. Individuals with clinically-significant coagulopathy at screening 36. Individuals with clinically-significant thrombocytopenia at screening 37. Hemoglobin < 12 g/dL at screening 38. Mean corpuscular volume (MCV) < 80 fL or > 100 fL at screening 39. Donation of whole blood within 8 weeks prior to the first experimental visit. Participation in the screening phase is permitted.

     40. History of inherent unremediable risks for anemia, such as hemoglobinopathies, hemolytic disorders, and bleeding disorders, regardless of whether their hemoglobin is currently normal.

     41. History of a large-volume gastrointestinal (GI) bleeding, such as a bleed that required ER evaluation or admission, required acute endoscopic or surgical management, was managed by blood transfusion, or caused anemia.

     42. History of NSAID-mediated peptic ulcer disease is excluded, irrespective of current medical treatment. A history of peptic ulcer disease from H. pylori does not exclude participation provided H. pylori was successfully eradicated. Other causes of peptic ulcer disease may be allowable, especially if definitively treated or the risk of recurrence is otherwise low.

     43. Chronic, untreated conditions that predispose to anemia, such as significant iron or B vitamin malabsorption, persistent menorrhagia, or other chronic or intermittent bleeding.

     44. Participation in an investigational drug study concurrently; participants who previously completed an investigational drug study cannot participate in the first experimental visit until at least 6 weeks after the final dose given during the previous investigational drug study. For the purposes of this exclusion, an investigational drug is a new chemical entity or a pharmaceutical investigated to support an initial new drug application. Furthermore, herbal or other supplements already deemed "generally regarded as safe" or legally sold in the U.S. would not be considered an investigational drug.

     45. Use of medications indicated for the treatment of diabetes within 6 weeks of the first experimental visit 46. Daily therapy with non-statin lipid-altering medications within 6 weeks of the first experimental visit is exclusionary, including long-term therapy with the agents listed below. Subjects may wash off these medications so long as the first experimental visit occurs at least 6 weeks after chronic therapy ceases. Following a washout period, fasting lipids will be repeated prior to the first experimental visit to assure that these are not exclusionary as defined above.
     1. Niacin > 100 mg/ day: (Niacor®, Slo-Niacin®, Niaspan®, Advicor®, Simcor®, Inositol Hexanicotinate, or supplemental niacin).
     2. Fibrates: gemfibrozil (Lopid®), fenofibrate (Antara®, Lofibra®, Tricor®, Triglide®), fenofibric acid (Trilipix®, Certriad®).
     3. Enterically active lipid altering drugs: colestipol (Colestid®), cholestyramine (Questran®), colesevelam (Welchol®), ezetimibe (Zetia®, Vytorin®), orlistat (Xenical®, Ali®).
     4. Prescription fish oil: Vascepa®, Epanova®, Lovaza® (nee Omacor®)
     5. Supplemental omega-3-enriched oils: flaxseed, fish, or algal oils
     6. Foods enriched with omega-3 fatty acids
     7. Consumption of up to 2 servings per week of fish is acceptable 47. Lipid-altering supplements

     <!-- -->

     1. Sterol/stanol products (e.g. CholestOff), policosanols
     2. Dietary fiber supplements, including >2 teaspoons of Metamucil® or psyllium containing supplements per day
     3. Garlic supplements or soy isoflavones supplements
     4. Supplemental vitamin B5 or related compounds unless part of a multi-vitamin
     5. As above, red yeast statin will be switched to a GMP prescription statin
     6. Any other medications, herbal products, or dietary supplements with known or potential lipid-altering effects 48. Anticoagulant therapy (except aspirin)

     <!-- -->

     1. Warfarin
     2. Rivaroxiban
     3. Apixaba
     4. Dabigantran 49. Anti-obesity medications or their components

     <!-- -->

     1. Orlistat (Xenical)
     2. Lorcaserin (Belviq)
     3. Phentermine plus extended-release topiramate (Qsymia)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Millar, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman School of Medicine at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Statin treated Caucasian adults with hypertriglyceridemia
Period: Overall Study
Arm/Group | Icosapent Ethyl | Usual Care
Started | 12 | 8
Baseline | 12 | 8
Treatment Visit (12 Week) | 11 | 7
Completed | 11 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unwilling to undergo required study procedure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Icosapent Ethyl | Usual Care | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
VLDL apoB100 Production Rate [Mean (Standard Deviation); unit: mg VLDL apoB100 / kg body weight per day] | 21.7 (10.8) | 14.9 (3.4) | 19.1 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in VLDL-apoB100 Production Rate
Description: The production rate of very low-density lipoprotein apolipoprotein B100 as determined by stable-isotope lipid kinetics techniques based on a primed constant infusion of deuterated leucine.
Time Frame: ≥ 13 weeks of observation on randomized treatment assignment
Population: All subjects who completed the ≥ 13 week treatment phase of the study (13-18 weeks).
Measure: Mean (Standard Deviation); unit: mg VLDL apoB100 / kg body weight per day
Arm/Group | Icosapent Ethyl | Usual Care
Number analyzed (Participants) | 11 | 7
mg VLDL apoB100 / kg body weight per day
  L apoB100 Production Rate (Baseline) | 21.7 (10.8) | 14.9 (3.4)
  VLDL apoB100 Production Rate (Treatment) | 21.3 (10.8) | 17.2 (8.5)
Statistical Analysis 1: Comparison: Icosapent Ethyl vs Usual Care; Test type: Superiority; p = 0.65, mixed effects regression; testing for the outcome employed mixed effects regression. The key fixed effects were group assignment, period, and the group X period interaction

ADVERSE EVENTS:
Time Frame: 12 weeks after subjects received their first daily dose of study drug or usual care.
Description: Adverse events were reported during scheduled visits during and after the 12 week treatment period.
Arm/Group | Icosapent Ethyl | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 8/12 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icosapent Ethyl (N=12) | Usual Care (N=8)
Constipation; Dyspepsia; Nausea; Gastroenteritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Headache; Migrane; Dizziness (Nervous system disorders) | 2 (2) | 5 (8)
Sinusitis; Itchy Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Limb discomfort; Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dermatitis; Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03885661/Prot_SAP_000.pdf